CLINICAL TRIAL: NCT02428725
Title: Platelet Reactivity Inhibition Following Ticagrelor Loading Dose and One Year Outcome in Patients Undergoing Percutaneous Coronary Intervention for an Acute Coronary Syndrome
Brief Title: Platelet Reactivity Inhibition Following Ticagrelor Loading Dose and One Year Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-A01913-44
Record Dates: First submitted 2015-03-26; First posted 2015-04-29 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute coronary syndrome patient (Experimental): Acute coronary syndrome patient undergoing PCI and eligible for ticagrelor therapy according to the guidelines accepting blood samples measuring platelets reactivity
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — Biological samples will be done to determine platelet reactivity testing by VASP-index, will be obtained between 6 and 12 hours after receiving ticagrelor

SUMMARY:
This study will try to determine if the measure of the platelet reactivity of the patients receiving from the ticagrelor continuation in an acute coronary syndrome handled by coronary angioplasty allows to predict the hemorrhagic risk.

DETAILED DESCRIPTION:
The use of thienopyridines in patients undergoing percutaneous coronary intervention (PCI) has dramatically decreased the rate of early stent thrombosis. Further the CURE trial demonstrated that long-term clopidogrel decreases the rate of major adverse cardiovascular events in acute coronary syndrome patients (ACS) . However clopidogrel has several limitations including a long delay of action which is a potential limitation in acute settings of coronary artery disease. Another major limitation of the drug is the wide inter individual variability in clopidogrel responsiveness related to various factors.

In addition recent studies suggested that platelet reactivity inhibition does also determine the bleeding risk.

The ticagrelor is a new blocker of the receiver P2Y12 which distinguishes itself from the clopidogrel by a superior biological efficiency. This biological property was translated in the study PLATO, having compared it with the clopidogrel in the ACS, by a reduction of the risk thrombotique. The ticagrelor is thus recommended in first intention in this indication. There seems be a variability of answer to the ticagrelor. Besides the ticagrelor infers a level of intense platelet inhibition which could explain on hemorrhagic risk which is associated with it.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome patient undergoing PCI and eligible for ticagrelor therapy according to the guidelines.

Exclusion criteria:

* New York Heart Association functional class III or IV
* Cardiac arrest
* Contra-indications to antiplatelet therapy
* Platelet count <100 G/l
* History of bleeding diathesis
* Concurrent severe illness with expected survival of < 1 year month
* Pregnant of childbearing woman
* Inability to provide an informed consent
* Contra indication to ticagrelor.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity inhibition measured by the VASP index 6 to 12 hours after the loading dose of ticagrelor | one year
  Platelet reactivity inhibition measured by the VASP index 6 to 12 hours after the loading dose is associated with the occurrence of BARC bleedings ≥ 2 at one year post-PCI.

SECONDARY OUTCOMES:
Relationship between VASP index and MACE | 1 month
  the rate of major cardiovascular events ( MACE )
Relationship between VASP index and MACE | 1 year
Relationship between VASP index and BARC | 1month
  BARC: bleeding academic research complications
Compliance to ticagrelor | 1 year
Evaluate Adenosine deaminase | 1 year
evaluate DDP IV activity | 1 year
Evaluate microparticules number and activity under ticagrelor | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BONELLO, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Laine M, Frere C, Cuisset T, Paganelli F, Morange PE, Dignat-George F, Berbis J, Camoin-Jau L, Bonello L. Potential mechanism of acute stent thrombosis with bivalirudin following percutaneous coronary intervention in acute coronary syndromes. Int J Cardiol. 2016 Oct 1;220:496-500. doi: 10.1016/j.ijcard.2016.06.247. Epub 2016 Jun 28. PMID 27390976